CLINICAL TRIAL: NCT03656094
Title: Chemotherapy Plus Pembrolizumab After Progression With Previous PD-1/PD-L1 Inhibitors in Patients With Advanced Non-small Cell Lung Cancer: Placebo-controlled Randomized Phase II Study
Brief Title: Chemotherapy With Pembrolizumab Continuation After Progression to PD-1/L1 Inhibitors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Mu Sun, Associate professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMC 2018-07-044
Record Dates: First submitted 2018-07-26; First posted 2018-09-04 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — pembrolizumab; Drug Therapy; Pemetrexed; Vinorelbine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab plus chemotherapy (Experimental): Pembrolizumab (200 mg) plus chemotherapy (physicians' choice among docetaxel, pemetrexed, or vinorelbine) every 3 weeks
  Interventions: Drug: Pembrolizumab plus chemotherapy
- Placebo plus chemotherapy (Active Comparator): Placebo plus chemotherapy (physicians' choice among docetaxel, pemetrexed, or vinorelbine) every 3 weeks
  Interventions: Drug: Placebo plus chemotherapy

INTERVENTIONS:
Drug: Pembrolizumab plus chemotherapy — Pembrolizumab plus chemotherapy
  Other Names: Chemotherapy: one of docetaxel, pemetrexed, or vinorelbine
  Arms: Pembrolizumab plus chemotherapy
Drug: Placebo plus chemotherapy — Placebo plus chemotherapy
  Other Names: chemotherapy: one of docetaxel, pemetrexed, or vinorelbine
  Arms: Placebo plus chemotherapy

SUMMARY:
After progression to previous PD-1/L1 inhibitors (pembrolizumab, nivolumab, or atezolizumab), physicians' choice chemotherapy plus pembolizumab (or placebo) will be administered (3 weeks per cycle) until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
Previous PD-1/PD-L1 inhibitors should be 2nd or 3rd line therapy for advanced NSCLC. There should be no systemic therapy after previous PD-1/PD-L1 therapy, before the enrollment to this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male /female participants who are at least 20 years of age on the day of signing informed consent with histologically confirmed diagnosis of
2. Histologically confirmed non-small cell carcinoma
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization.
4. Received one or two cytotoxic chemotherapy for advanced NSCLC including at least one platinum-doublet
5. Has received prior therapy with an anti-PD-1, anti-PD-L1 agents (monotherapy) and progression to last PD-1/PD-L1 inhibitors. The last PD-1/PD-L1 inhibitor should be administered 6 weeks before the study enrollment, and no other systemic therapy should be done between the interval.
6. At least one measurable lesion Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Available data for PD-L1 IHC results (any of one tested by 22C3, SP263, or SP142) irrespective of expression level.
8. EGFR and ALK wild type

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to [randomization/allocation] (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior systemic anti-cancer therapy including investigational agents within 3 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to [randomization /allocation].

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
3. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
4. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 3 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, well differentiated thyroid carcinoma, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
8. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment. Patients with oligo (≤5) brain metastasis with size less than 1cm can be enrolled without prior radiotherapy, if the tumors are regarded as asymptomatic and stable, based on follow-up brain MRIs checked intervals of at least 3 months. However, all patients with previously non-irradiated brain metastases should have brain MRI checked within 4 weeks before starting administration of study drugs.
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any PD-1/PD-L1 inhibitors.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a known history of Human Immunodeficiency Virus (HIV)
14. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
15. Has a known history of active TB (Bacillus Tuberculosis).
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 60 moths
  Time interval from enrollment to disease progression or death

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 60 months
  Partial reseponse is defined as a decrease by 30% or more in sums of longest diameter of measurable target lesions
Overall survival (OS) | 60 months
  Time interval between enrollment to death of any cause
Toxicity by CTCAE | 60 months
  AEs graded using CTCAE (Version 4.0) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Mu Sun, Principal Investigator — Samsung Medical Center
Locations (1):
- Jong-Mu Sun, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No